CLINICAL TRIAL: NCT05494398
Title: Targeting the Neurobiology of Restricted and Repetitive Behaviors in Children With Autism Using N-acetylcysteine: an Open Label Extension
Brief Title: Targeting the Neurobiology of RRB in Autism Using N-acetylcysteine: Open Label
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, John Patrick Hegarty, Instructor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-64292; K99HD101702 (NIH)
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder
Keywords: Magnetic Resonance Imaging; N-acetylcysteine; Restricted and Repetitive Behaviors; Electroencephalography
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- N-Acetylcysteine (Experimental)
  Interventions: Drug: N-acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine — 12 week administration of N-Acetylcysteine to target restricted repetitive behavior severity.

SUMMARY:
The goal of this study is to target the neurobiology of restricted and repetitive behaviors in children with autism spectrum disorder using N-acetylcysteine (NAC), a well-tolerated nutritional supplement that has shown promise for reducing symptom severity in recent small-scale trials. The findings from this research will shed light on the mechanisms of action underlying the clinical benefits of NAC and the effects of NAC on altering restricted and repetitive behavior symptom severity in children with autism spectrum disorder.

ELIGIBILITY:
Inclusion Criteria:

* participation in an associated single-dose (IRB-54931, NCT04278898) or randomized, controlled trial of NAC (IRB- 68353, NCT05664789).
* stable medication regimens (≥ 30 days) with no anticipated changes during the trial.

Exclusion criteria:

• the presence of significant medical problems that reduce medical stability.

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in glutamatergic neurometabolites (Glx) measured by proton spectroscopy Magnetic Resonance Imaging (MRI) | Baseline and Week 12 of treatment
Change in restricted and repetitive behaviors as measured by Children's Yale Brown Obsessive Compulsive Scale - Autism Spectrum Disorder (CYBOCS-ASD) | Screening, Week 8, week 12
  Higher scores on the Children's Yale Brown Obsessive Compulsive Scale - Autism Spectrum Disorder mean higher levels of restricted and repetitive behaviors (Raw Score Total Range: 0-20)

SECONDARY OUTCOMES:
Change in Gamma band amplitude and synchronization measured by electroencephalography (EEG) | Baseline, Week 12
Change in restricted repetitive behavior subtypes as measured by the Restricted Behavior Scale - Revised (RBS-R) | Baseline, week 8, week 12
  Higher scores on the Repetitive Behavior Scale- Revised mean higher levels of repetitive and restricted behaviors. (Raw Score Total Range: 0 - 129)

CONTACTS AND LOCATIONS:
Overall Officials: John Hegarty, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-Identified data will be shared with the National Database for Autism Research (NDAR)
Time Frame: The data will be submitted on January 15th and July 15th each year.
Access Criteria: Researchers with access to the National Database for Autism Research (NDAR) will be able to obtain the submitted data
URL: http://nda.nih.gov